CLINICAL TRIAL: NCT06538116
Title: A Randomized, Double-Blinded Study to Evaluate the Efficacy and Safety of Mevidalen in Patients With Alzheimer's Disease
Brief Title: A Study of Mevidalen (LY3154207) in Participants With Alzheimer's Disease
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18822; I7S-MC-HBEO (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-08-01; First posted 2024-08-05 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — LY3154207

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Mevidalen (high dose) (Experimental): Mevidalen high dose administered orally.
  Interventions: Drug: Mevidalen
- Mevidalen (low dose) (Experimental): Mevidalen low dose administered orally.
  Interventions: Drug: Mevidalen
- Placebo (Placebo Comparator): Placebo administered orally.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mevidalen — Administered orally
  Other Names: LY3154207
  Arms: Mevidalen (high dose); Mevidalen (low dose)
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The main purpose of this study is to look at how safe the study drug (mevidalen) is and whether it works to alleviate symptoms when given to people with mild to moderate Alzheimer Disease (AD) dementia. This is done by looking at participants: thinking and memory (cognition), everyday activities and sleep, AD symptoms, physical activity, irritability or anxiety. The study is expected to last approximately 26 weeks and may include up to 14 visits.

ELIGIBILITY:
Inclusion Criteria:

* Have gradual and progressive decline in memory function for greater than or equal to 6 months that is severe enough to interfere with activities of daily living.
* Have MMSE score of 13 to 24.
* Have eligibile plasma P-tau or historical evidence of AD pathology.
* Have a reliable study partner who will provide written informed consent to participate, is in frequent contact with the participant and will be available at designated times.
* Males with partners of childbearing potential must agree to abide with provided contraception guidance.

Exclusion Criteria:

* Are individuals of childbearing potential.
* Have significant central nervous system or psychiatric disease, other than AD, that in the investigator's opinion may affect cognition or the ability to complete the study (e.g: head trauma, stroke, seizure disorder etc.,).
* Have cardiovascular-related risk factors or history that include uncontrolled hypertension, heart failure, stroke; or liver-related abnormalities.
* Use of moderate or strong CYP3A4 inhibitors or inducers.
* Have participated within the last 30 days in a clinical trial involving an investigational product.
* Participant is, in the judgment of the investigator, actively suicidal and therefore deemed to be at significant risk for suicide.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-08-26 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Integrated Alzheimer's Disease Rating Scale (iADRS) | Baseline, Week 24
  iADRS assesses the impact of cognitive loss on everyday activities and provides a measure of global AD severity as a single summary score. It comprises of 2 underlying domains "cognitive ability" and "functional ability," and integrates the items in both the domains a single overall score ranging from 0 to 144, with lower scores indicating worse performance.

SECONDARY OUTCOMES:
Change from Baseline in Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog13) | Baseline, Week 24
  The ADAS-Cog13 consists of 13 items which assess the areas of cognitive function that are the most typically impaired in AD: orientation, verbal memory, language, praxis, delayed free recall, and digit cancellation measures. The scale ranges from 0 to 85, with higher scores indicating greater disease severity.
Change from Baseline in Verbal Fluency Test | Baseline, Week 24
  The Verbal Fluency Test, also known as the FAS test, requires participants to say as many words as possible beginning with specific letters (F, A, and S) in 1 minute. The FAS score corresponds to the number of words generated by each participant under each letter category within 1 minute. A higher score indicates better performance.
Change from Baseline in Category Fluency Test | Baseline, Week 24
  The Category Fluency test is a measure of semantic memory and involves planning, organization, and cognitive flexibility. The participant is asked to generate as many words as possible in 1 minute that belong to the animal semantic category. Total score is the sum of correct words generated for the animal category, and higher values indicate better performance.
Change from Baseline in Digit Symbol Coding Test( Wechsler Adult Intelligence Scale-IV)(WAIS-IV) | Baseline, Week 24
  The Digit Symbol-Coding test from the WAIS-IV involves testing processing speed among subjects; The digit symbol coding requires a subject to match symbols to numbers according to a key. The number of correct symbols within the allowed time constitutes the score, and higher values indicate better performance.
Change from Baseline in Mini Mental State Examination (MMSE) | Baseline, Week 24
  The MMSE is a brief instrument used to assess global cognition. The instrument measures orientation, memory, attention, ability to name objects, follow verbal/written commands, write a sentence, and copy figures. Total score ranges from 0 to 30, with lower score indicating greater level of impairment.
Change from Baseline in Alzheimer's Disease Cooperative Study-Activities of Daily Living (ADCS-ADL) | Baseline, Week 24
  The ADCS-ADL is a 23-item inventory developed as a rater-administered questionnaire that is to be answered by the participant's study partner. Study partner is asked to observe and rate the performance of activities of daily living attempted by participants. The range for the total ADCS-ADL score is 0 to 78, with lower scores indicating greater level of impairment.
Alzheimer's Disease Cooperative Study-Clinical Global Impression of Change score (ADCS-CGIC) | Week 24
  The ADCS-CGIC is a 7-point, categorical scale that provides a single global rating of change from baseline. A score of 1 indicates marked improvement; a score of 2, moderate improvement; a score of 3, minimal improvement; a score of 4, no change; a score of 5, minimal worsening; a score of 6, moderate worsening; and a score of 7, marked worsening.
Change from Baseline on Neuropsychiatric Inventory (NPI-12) | Baseline, Week 24
  The NPI-12 is rating instrument to assess abnormal behaviors in dementia patients by informant-based interview that utilizes scripted questions to explore 12 different symptom domains: delusions, hallucinations, agitation/aggression, dysphoria, anxiety, euphoria, apathy, disinhibition, irritability/lability, aberrant motor activity, night-time behavioral disturbances, and appetite and eating abnormalities. The frequency of behaviour is scored from 0 (Rarely) to 4 (very often) and the severity from 0 (mild) to 3 (severe). A total score for each symptom is calculated by multiplying the frequency rating by the severity rating. The total NPI-12 score is the sum of all symptom scores and ranges from 0 to 144, with higher scores indicating a greater degree of symptomatology.
Change from Baseline on Epworth Sleepiness Scale (ESS) | Baseline, Week 24
  ESS is an 8-item questionnaire that measures the chances of "dozing off" in different daytime situations over the past week. Scores range from 0 to 24, with scores greater than or equal to 10 indicating excessive daytime sleepiness.
Change from Baseline on Quick Dementia Rating Scale (QDRS) | Baseline, Week 24
  The QDRS is a 10-item rating scale that assesses aspects of cognition, behavior, and daily functioning on a 5-point scale where no problems = 0, slight problems = 0.5, mild problems = 1, moderate to severe problems = 2, and severe problems = 3. Total scores range from 0 to 30 and higher scores indicate increased cognitive impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (64):
- United States (44):
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Baptist Health Center for Clinical Research LLC, Little Rock, Arkansas
  - Profound Research LLC At The Neurology Center of Southern California, Carlsbad, California
  - Neuropain Medical Center, Fresno, California
  - Catalina Research Institute, Montclair, California
  - California Neuroscience Research, LLC, Sherman Oaks, California
  - JEM Research Institute, Atlantis, Florida
  - Visionary Investigators Network, Aventura, Florida
  - Excel Medical Clinical Trials, LLC Boca Raton dba Flourish Research, Boca Raton, Florida
  - Vertex Clinical Research, Clermont, Florida
  - Neuropsychiatric Research Center of Southwest Florida, Fort Myers, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Merritt Island Medical Research, LLC dba Flourish Research, Merritt Island, Florida
  - Visionary Investigators Network, Miami, Florida
  - Suncoast Clinical Research - New Port Richey, New Port Richey, Florida
  - Renstar Medical Research, Ocala, Florida
  - Charter Research, LLC, Orlando, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Intercoastal Medical Group, Sarasota, Florida
  - Brain Matters Research, Stuart, Florida
  - Charter Research - The Villages, The Villages, Florida
  - Premiere Research Institute at Palm Beach Neurology, West Palm Beach, Florida
  - Conquest Research, Winter Park, Florida
  - Accel Research Sites - NeuroStudies CRU, Decatur, Georgia
  - CenExel iResearch Atlanta, Decatur, Georgia
  - CenExel iResearch, LLC, Savannah, Georgia
  - Hawaii Pacific Neuroscience, Honolulu, Hawaii
  - Ascension Alexian Brothers, Elk Grove Village, Illinois
  - Josephson, Wallack, Munshower Neurology, P.C., Indianapolis, Indiana
  - ActivMed Practices & Research, LLC, Methuen, Massachusetts
  - QUEST Research Institute, Farmington Hills, Michigan
  - CenExel Advanced Memory Research Institute of NJ, Toms River, New Jersey
  - AMC Research, LLC dba Flourish Research, Matthews, North Carolina
  - Eximia Clinical Research-NC, LLC, Raleigh, North Carolina
  - Keystone Clinical Studies, LLC Philadelphia dba Flourish Research, Plymouth Meeting, Pennsylvania
  - Clinical Neuroscience Solutions, Inc.Ta, Memphis, Tennessee
  - Senior Adults Specialty Research, Austin, Texas
  - Kerwin Medical Center, Dallas, Texas
  - Cedar Health Research, LLC, Euless, Texas
  - Clinical Trial Network LLC, Houston, Texas
  - El Faro Health and Therapeutics, Rio Grande City, Texas
  - Be Well Clinical Studies, Round Rock, Texas
  - Clinical Trials of Texas, LLC San Antonio dba Flourish Research, San Antonio, Texas
  - University of Washington Medical Center, Seattle, Washington
- Japan (20):
  - Akita City Hospital, Akita
  - Memory Clinic Ochanomizu, Bunkyō City
  - Inage Neurology and Memory Clinic, Chiba
  - Ikuseikai Shinozuka Hospital, Fujioka-shi
  - Mental Clinic Sakurazaka, Fukuoka
  - Kuramitsu Hospital, Fukuoka
  - Himeji Central Hospital Clinic, Himeji-shi
  - Koseikai Cocoro Hospital Kusatsu, Hiroshima
  - NHO Hizen Psychiatric Medical Center, Kanzaki-gun
  - Rainbow & Sea Hospital, Karatsu-shi
  - Kishikai Kishi Hospital, Kiryu-shi
  - Southern TOHOKU Medical Clinic, Koriyama-shi
  - Katayama Medical Clinic, Kurashiki-shi
  - Mabashi Clinic, Matsudo-shi
  - National Center for Geriatrics and Gerontology, Obu-shi
  - Tokyo Medical University Hospital, Shinjuku-ku
  - Tokyo Metropolitan Bokutoh Hospital, Sumida-ku
  - Memory Clinic Toride, Toride-shi
  - Yamagata University Hospital, Yamagata
  - Oita University Hospital, Yufu-shi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of Mevidalen (LY3154207) in Participants With Alzheimer's Disease — https://trials.lilly.com/en-US/trial/524115